CLINICAL TRIAL: NCT04912622
Title: Cross Sectional Study: in Vivo Morphometric Characterisation of Human Retinal Pigment Epithelium With Transscleral Optical Phase Imaging in Photoreceptor/ Retinal Pigment Epithelium/ Bruch's Membrane/ Choriocapillaris Complex Disorders
Brief Title: RPE Characterisation With Transscleral Optical Phase Imaging in Retinal Disorders
Acronym: CEL01LUKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Cellularis Studie 01; EKNZ2020-02454 (Other: BASEC)
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Retinal Disease; Eye Disease
MeSH Terms: conditions — Retinal Diseases; Eye Diseases

STUDY DESIGN:
Intervention Model Description: Control group: 110 individuals with healthy retina Patient group: 95 individuals with diseased retina Exclusion: age < 18y, pregnancy, epilepsy, no informed consent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Device: Cellularis version 2.0 imaging Image acquisition of retinal pigment epithelium (RPE) cells of central retina with consecutive qualitative and quantitative description of these retinal cell layers.
  Interventions: Diagnostic Test: Clinical Trial
- Patient (Experimental): Device: Cellularis version 2.0 imaging Image acquisition of retinal pigment epithelium (RPE) cells of central retina with consecutive qualitative and quantitative description of these retinal cell layers.
  Interventions: Diagnostic Test: Clinical Trial

INTERVENTIONS:
Diagnostic Test: Clinical Trial — Retinal image acquisition with Cellularis version 2.0

SUMMARY:
Accumulating evidence suggest that the functional unit of photoreceptor/ retinal pigment epithelium (RPE)/Bruch's membrane/choriocapillaris plays a key role in pathophysiologic processes of a wide range of medical retinal disorders of the eye. Little is known about in vivo morphometric characteristics of human RPE cells as in vivo observation of these cells was so far technically challenging and hence nearly impossible to implement in a clinical setting. Transscleral optical phase imaging is a novel in-vivo microscopy technique allowing human RPE imaging on a cellular level with the potential of clinical application in a multimodal retinal imaging approach for diagnostic purpose in medical retina patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Patients with a medical retinal disease involving the retinal pigment epithelium (age related macular degeneration, diabetic retinopathy, retinal vascular occlusive disease, central serous chorioretinopathy, tapetoretinal degeneration)
* Participants with healthy eyes for the control group

Exclusion Criteria:

* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia etc. of the participant
* Aged < 18 years.
* Pregnancy
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
RPE morphology | 12 months
  RPE cell density (number of cells per mm^2)

SECONDARY OUTCOMES:
averaged RPE cell area [um2] Averaged number of neighbors of RPE cells [unitless] Averaged RPE spacing [um] Averaged RPE pigmentation parameter [unitless] | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Luzern, Lucerne, Switzerland